CLINICAL TRIAL: NCT02404441
Title: Open Label Multicenter Phase I/II Study of the Safety and Efficacy of PDR001 Administered to Patients With Advanced Malignancies
Brief Title: Phase I/II Study of PDR001 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001X2101; 2014-003929-17 (EudraCT Number)
Record Dates: First submitted 2015-03-20; First posted 2015-03-31 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Melanoma; Non-small Sell Lung Cancer (NSCLC); Triple Negative Breast Cancer; Anaplastic Thyroid Cancer; Other Solid Tumors
Keywords: Phase I/II; PDR001; Checkpoint inhibitor; PD-1; PD-L1; NSCLC
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Thyroid Carcinoma, Anaplastic | interventions — spartalizumab

STUDY DESIGN:
Intervention Model Description: Although the study had 2 'arms', the phase I part of the study had 5 dosing cohorts and the phase ll part had 5 treatment groups for a total of 10 reporting groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- patients with solid tumors (Other): Phase I Dose escalation cohorts
  Interventions: Biological: PDR001
- Selected tumor types (Other): Phase II expansion: Selected tumor types: melanoma, NSCLC, triple negative breast cancer, anaplastic thyroid cancer
  Interventions: Biological: PDR001

INTERVENTIONS:
Biological: PDR001 — anti-PD1 antibody

SUMMARY:
The purpose of this "first-in-human" study of PDR001 was to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and antitumor activity of PDR001 administered i.v. as a single agent to adult patients with solid tumors.

By blocking the interaction between PD-1 and its ligands, PD-L1 and PD-L2, PDR001 inhibits the PD-1 immune checkpoint, resulting in activation of an antitumor immune response by activating effector T-cells and inhibiting regulatory T-cells.

DETAILED DESCRIPTION:
This study was designed as a phase I/II, multi-center, open-label study starting with a phase I dose escalation part followed by a phase II part.

Although the study had 2 'arms', the phase I part of the study had 5 dosing cohorts and the phase ll part had 5 treatment groups for a total of 10 reporting groups.

PDR001 was administered every 2 weeks until patient experienced unacceptable toxicity, progressive disease per immune related Response Criteria (irRC) and/or treatment was discontinued at the discretion of the investigator or the patient.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must have been obtained prior to any screening procedures
* Phase I part: Patients with advanced/metastatic solid tumors, with measurable or non-measurable disease as determined by RECIST version 1.1 (refer to Appendix 1), who have progressed despite standard therapy or are intolerant of standard therapy, or for whom no standard therapy exists.
* Phase II part: Patients with advanced/metastatic solid tumors, with at least one measurable lesion as determined by RECIST version 1.1, who have progressed following their last prior therapy, and fit into one of the following groups:

  * Group 1a and 1b: NSCLC:

Patients with NSCLC must have had disease recurrence or progression during or after no more than one prior systemic chemotherapy regimen (platinum doublet-based) for advanced or metastatic disease. Prior maintenance therapy is allowed (e.g. pemetrexed, erlotinib, bevacizumab).

Only patients with EGFR mutation-negative tumor are eligible (defined as negative for exon 19 deletions and for the L858R mutation in EGFR at a minimum; however, if more extensive EGFR mutation testing has been performed, the tumor must not harbor any known activating EGFR mutations in Exons 18-21 in order to be considered EGFR mutation-negative). All patients must be tested for EGFR mutational status and, for ALK translocation status if no mutation is detected in EGFR. Patients with ALK translocation-positive NSCLC must have had disease progression following treatment with a corresponding inhibitor and no more than one systemic chemotherapy regimen (platinum doublet-based), in any sequence.

* Group 2: Melanoma:

All patients must have been tested for BRAF mutations. Patients with V600 mutation positive melanoma must have clinical or radiological evidence of disease progression during or after treatment with a BRAF inhibitor alone or in combination with other agents.

* Group 3: Triple negatice breast cancer.
* Group 4: Anaplastic thyroid cancer
* Patients are not required to have received or progressed on a prior therapy.
* Patients must not be at short term risk for life threatening complications (such as airway compromise or bleeding from locoregional or metastatic disease).
* Chemoradiation and/or surgery should be considered prior to study entry for those patients with locally advanced disease if those therapies are considered to be in the best interest of the patient.

  * ECOG Performance Status ≤ 1.
  * Patients must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy. Patient must be willing to undergo a new tumor biopsy at baseline or at molecular pre-screening if applicable, and during therapy on this study. For patients in the phase II part of the study, exceptions may be granted after documented discussion with Novartis. After a sufficient number of paired biopsies are collected, the decision may be taken to stop the collection of biopsies.

Exclusion Criteria:

* History of severe hypersensitivity reactions to other mAbs
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Active infection requiring systemic antibiotic therapy.
* HIV infection.
* Active HBV or HCV infection.
* Patients with ocular melanoma.
* Systemic anti-cancer therapy within 2 weeks of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity, e.g. mitomycin C and nitrosoureas, 4 weeks washout period. For patients receiving anticancer immunotherapies such as CTLA-4 antagonists, 6 weeks is indicated as the washout period.
* Prior PD-1- or PD-L1-directed therapy.
* Patients requiring chronic treatment with systemic steroid therapy, other than replacement-dose steroids in the setting of adrenal insufficiency. Topical, inhaled, nasal and ophthalmic steroids are not prohibited.
* Patients receiving systemic treatment with any immunosuppressive medication (other than steroids as described above).
* Use of any vaccines against infectious diseases (e.g. influenza, varicella, pneumococcus) within 4 weeks of initiation of study treatment.
* Presence of ≥ CTCAE grade 2 toxicity (except alopecia, peripheral neuropathy and ototoxicity, which are excluded if ≥ CTCAE grade 3) due to prior cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- United States (6):
  - The Sidney Kimmel Cancer Center at Johns Hopkins Hospital Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Oregon Health and Science University SC-10, Portland, Oregon
  - Sarah Cannon Research Institute SCRI RC, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center MD Anderson PSC, Houston, Texas
  - Huntsman Cancer Institute Univ. of Utah HCI, Salt Lake City, Utah
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (3):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Ulm
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, El Achrafiyé, Lebanon
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leiden
- Novartis Investigative Site, Oslo, Norway
- Poland (4):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Edirne
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Capdevila J, Wirth LJ, Ernst T, Ponce Aix S, Lin CC, Ramlau R, Butler MO, Delord JP, Gelderblom H, Ascierto PA, Fasolo A, Fuhrer D, Hutter-Kronke ML, Forde PM, Wrona A, Santoro A, Sadow PM, Szpakowski S, Wu H, Bostel G, Faris J, Cameron S, Varga A, Taylor M. PD-1 Blockade in Anaplastic Thyroid Carcinoma. J Clin Oncol. 2020 Aug 10;38(23):2620-2627. doi: 10.1200/JCO.19.02727. Epub 2020 May 4. PMID 32364844
- [Derived] Naing A, Gainor JF, Gelderblom H, Forde PM, Butler MO, Lin CC, Sharma S, Ochoa de Olza M, Varga A, Taylor M, Schellens JHM, Wu H, Sun H, Silva AP, Faris J, Mataraza J, Cameron S, Bauer TM. A first-in-human phase 1 dose escalation study of spartalizumab (PDR001), an anti-PD-1 antibody, in patients with advanced solid tumors. J Immunother Cancer. 2020 Mar;8(1):e000530. doi: 10.1136/jitc-2020-000530. PMID 32179633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 patients were analyzed in Phase l and 261 patients were analyzed in Phase II of this study.
Pre-assignment Details: The study planned to analyze about 58 patients in Phase I and about 120 patients in Phase II.
Groups:
- 1mg/kg q2w: Phase I Dose escalation cohort patients who took PDR001 1 mg/kg q2w
- 3mg/kg q2w: Phase I Dose escalation cohort patients who took PRD001 3 mg/kg q2w
- 10mg/kg q2w: Phase I Dose escalation cohort patients who took PRD001 10 mg/kg q2w
- 3mg/kg q4w: Phase I Dose escalation cohort patients who took PRD001 3 mg/kg q4w
- 5mg/kg q4w: Phase I Dose escalation cohort patients who took PRD001 5 mg/kg q4w
- NSCLC 400mg/q4w: Phase II: non-small cell cancer patients who took PDR001 400 mg/q4w
- Melanoma 400mg/q4w: Phase II: Melanoma patients who took PDR001 400 mg/q4w
- TNBC 400mg/q4w: Phase II: Triple negative breast cancer (TNBC) patients who took PDR001 400 mg/q4w
- NSCLC 300mg/q3w: Phase II: non-small cell cancer patients who took PDR001 300 mg/q3w
- ATC 400 mg/q4w: Patients in Phase II with anaplastic thyroid cancer (ATC) who took PDR001 400 mg/q4w
Period: Phase 1 Part
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w | NSCLC 400mg/q4w | Melanoma 400mg/q4w | TNBC 400mg/q4w | NSCLC 300mg/q3w | ATC 400 mg/q4w
Started | 16 | 15 | 11 | 6 | 10 | 0 | 0 | 0 | 0 | 0
Completed (Completed = Treatment Discontinued) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 15 | 11 | 6 | 10 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 14 | 11 | 7 | 6 | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Subject/Guardian Decision | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 Part
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w | NSCLC 400mg/q4w | Melanoma 400mg/q4w | TNBC 400mg/q4w | NSCLC 300mg/q3w | ATC 400 mg/q4w
Started | 0 | 0 | 0 | 0 | 0 | 59 | 61 | 40 | 59 | 42
Entered Post-treatment Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 1 | 6 | 1
No Longer Being Followed for Post-treatment Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 1 | 6 | 1
Entered Survival Follow-up | 0 | 0 | 0 | 0 | 0 | 38 | 34 | 26 | 35 | 25
Completed (Completed = Treatment Discontinued) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 59 | 61 | 40 | 59 | 42
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 6 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 7 | 9 | 2 | 1 | 3
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 43 | 32 | 31 | 39 | 27
Not completed — Subject/guardian decision | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 0 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 4 | 10 | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS included all subjects who received at least one dose of spartalizumab. Subjects were analyzed according to the planned treatment (dose level and regimen).
Groups:
- 10mg/kg q2w: Phase I Dose escalation cohort patients who took PDR001 10 mg/kg q2w
- Total: Total of all reporting groups
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w | NSCLC 400mg/q4w | Melanoma 400mg/q4w | TNBC 400mg/q4w | NSCLC 300mg/q3w | ATC 400 mg/q4w | Total
Number analyzed (Participants) | 16 | 15 | 11 | 6 | 10 | 59 | 61 | 40 | 59 | 42 | 319
Age, Customized [Number; unit: Participants]
  < 65 years | 12 | 9 | 8 | 6 | 8 | 33 | 37 | 29 | 35 | 25 | 202
  ≥ 65years | 4 | 6 | 3 | 0 | 2 | 26 | 24 | 11 | 24 | 17 | 117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 4 | 2 | 4 | 23 | 22 | 40 | 20 | 19 | 150
  Male | 7 | 8 | 7 | 4 | 6 | 36 | 39 | 0 | 39 | 23 | 169
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 10 | 14 | 8 | 4 | 8 | 42 | 37 | 32 | 50 | 33 | 238
  Black | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 5
  Asian | 3 | 1 | 2 | 2 | 1 | 12 | 23 | 4 | 8 | 4 | 60
  Unknown | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 1 | 4 | 13
  Other | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase l: The Exposure (AUC(0-336h)) After First Dose of Treatment at Cycle 3 (Each Cycle = 28 Days)
Description: Estimated the recommended phase 2 dose (RP2D) and/or the maximum tolerated dose (MTD) for PDR001.
  AUC0-336h is the AUC from time zero to 336 hour post dose of a measurable concentration sampling time.
Time Frame: Predose, 1hour (h), 24h, 48h, 72h, 168h, 240h, 336h post dose (cycle 3)
Population: Pharmacokinetic analysis set (PAS): The PAS consisted of all subjects who had at least one blood sample providing evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w
Number analyzed (Participants) | 8 | 4 | 4 | 3 | 4
day*ug/mL | 270 (52.5) | 1150 (51.1) | 3110 (33.1) | 575 (21.8) | 1490 (34.2)

2. Primary Outcome: Phase l: Incidence of Dose Limiting Toxicities (DLTs)
Description: DLT is defined as an adverse event (AE) or abnormal laboratory value of common terminology criteria for adverse events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications, which occurs within the first cycle of treatment with PDR001 during the dose escalation part of the study for which relationship to study treatment cannot be ruled out, with some exceptions.
Time Frame: 8 months
Population: Safety Set: The Safety Set included all subjects from the FAS who received at least one dose of spartalizumab and had at least one valid post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w
Number analyzed (Participants) | 16 | 15 | 11 | 6 | 10
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase ll: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Description: ORR is the percentage of participants with a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 CR = at least 2 determinations of CR at least 4 weeks apart before progression where confirmation required or 1 determination of CR prior to progression where confirmation not required.
  PR = at least 2 determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) where confirmation required or 1 determination of PR prior to progression where confirmation not required.
  RECIST criteria is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
Time Frame: 61 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- NSCLC 400 mg/q4w: Patients in Phase II with non-small cell cancer who took PDR001 400 mg/q4w
- Melanoma 400 mg/q4w: Patients in Phase II with Melanoma who took PDR001 400 mg/q4w
- TNBC 400 mg/q4w: Patients in Phase II with TNBC who took PDR001 400 mg/q4w
- NSCLC 300 mg/q3w: Patients in Phase II with non-small cell cancer who took PDR001 300 mg/q3w
- All Phase II Patients: All patients in Phase II regardless of how they took PDR001
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w | All Phase II Patients
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42 | 261
Percentage of participants | 15.3 [8.2 to 25.1] | 27.9 [18.6 to 38.8] | 0.0 [0.0 to 7.2] | 6.8 [2.3 to 14.8] | 19.0 [9.8 to 31.8] | 14.6 [11.1 to 18.6]

4. Secondary Outcome: Phase I: Serum Pharmacokinetic (PK) Parameter AUCs (AUC0-336h (Cycle 1 Only), AUCinf, AUClast AUCtau)
Description: AUC0-336h is the AUC from time zero to 336 hour post dose of a measurable concentration sampling time.
  AUClast: The AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1).
  AUCinf: The AUC from time zero to infinity (mass x time x volume-1). AUCtau: The AUC calculated to the end of a dosing interval (tau) at steady-state (amount x time x volume-1).
Time Frame: Predose, 1hour (h), 24h, 48h, 72h, 168h, 240h, 336h post dose (cycle 1 & 3)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w
Number analyzed (Participants) | 16 | 15 | 11 | 6 | 10
day*ug/mL
  Cycle (C) 1: AUC0-336h (n=16, 13, 10, 6, 10): number analyzed (Participants) | 16 | 13 | 10 | 6 | 10
  Cycle (C) 1: AUC0-336h (n=16, 13, 10, 6, 10) | 126 (29.5) | 324 (24.4) | 1270 (20.3) | 350 (35.0) | 638 (35.3)
  C1: AUCinf (n = 1, 0,0,2,3): number analyzed (Participants) | 1 | 0 | 0 | 2 | 3
  C1: AUCinf (n = 1, 0,0,2,3) | 123 (0) |  |  | 384 (9.8) | 726 (16.0)
  C1: AUClast | 125 (29.9) | 353 (31.4) | 1240 (21.6) | 522 (39.1) | 943 (37.4)
  C1: AUCtau (n = 16, 13, 10, 6, 10): number analyzed (Participants) | 16 | 13 | 10 | 6 | 10
  C1: AUCtau (n = 16, 13, 10, 6, 10) | 126 (29.5) | 324 (24.4) | 1270 (20.3) | 524 (39.6) | 984 (41.9)
  C3: AUClast: number analyzed (Participants) | 11 | 9 | 5 | 3 | 4
  C3: AUClast | 260 (44.8) | 995 (60.5) | 2520 (58.4) | 933 (21.3) | 2560 (37.2)
  C3: AUCtau (n = 8, 4, 4, 2, 2): number analyzed (Participants) | 8 | 4 | 4 | 2 | 2
  C3: AUCtau (n = 8, 4, 4, 2, 2) | 270 (52.5) | 1150 (51.1) | 3110 (33.1) | 1040 (19.1) | 2770 (26.6)

5. Secondary Outcome: Phase I: Serum Pharmacokinetic (PK) Parameter Cmax
Description: The maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass x volume-1)
Time Frame: Predose, 1hour (h), 24h, 48h, 72h, 168h, 240h, 336h post dose (Cycle 1 & 3)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w
Number analyzed (Participants) | 16 | 15 | 11 | 6 | 10
ug/mL
  C1 (n = 15, 15, 10, 6, 9): number analyzed (Participants) | 15 | 15 | 10 | 6 | 9
  C1 (n = 15, 15, 10, 6, 9) | 18.2 (26.5) | 53.8 (23.6) | 185 (18.3) | 53.8 (29.4) | 106 (34.2)
  C3 (n = 10, 7, 3, 3, 2): number analyzed (Participants) | 10 | 7 | 3 | 3 | 2
  C3 (n = 10, 7, 3, 3, 2) | 29.7 (41.0) | 112 (27.3) | 312 (30.0) | 69.7 (9.4) | 179 (45.2)

6. Secondary Outcome: Phase I: Serum Pharmacokinetic (PK) Parameter Tmax
Description: The time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration (time)
Time Frame: Predose, 1hour (h), 24h, 48h, 72h, 168h, 240h, 336h post dose (cycle 1 & 3)
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w
Number analyzed (Participants) | 16 | 15 | 11 | 6 | 10
hour
  C1 (n = 15, 15, 10, 6, 9): number analyzed (Participants) | 15 | 15 | 10 | 6 | 9
  C1 (n = 15, 15, 10, 6, 9) | 1.58 [1.38 to 2.12] | 1.57 [1.25 to 1.7] | 1.55 [1.13 to 1.68] | 1.55 [1.5 to 1.83] | 1.58 [1.08 to 1.67]
  C3 (n = 10, 7, 3, 3, 2): number analyzed (Participants) | 10 | 7 | 3 | 3 | 2
  C3 (n = 10, 7, 3, 3, 2) | 1.55 [1.45 to 1.75] | 1.55 [0.75 to 1.58] | 1.58 [1.52 to 1.62] | 1.5 [1.5 to 1.57] | 1.3 [0.783 to 1.82]

7. Secondary Outcome: Phase ll: Serum Pharmacokinetic (PK) Parameter AUCs (AUC336h, AUCinf, AUClast, AUCtau)
Description: as for outcome 4
Time Frame: Predose, 1hour (h), 24h, 48h, 72h, 168h, 240h, 336h post dose (cycle 1 & 3)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42
day*ug/mL
  C1: AUC0-336h (n =58, 58, 37, 54, 37): number analyzed (Participants) | 58 | 58 | 37 | 54 | 37
  C1: AUC0-336h (n =58, 58, 37, 54, 37) | 681 (39.4) | 775 (31.7) | 752 (29.3) | 535 (38.3) | 704 (28.2)
  C1: AUCinf (n = 13, 8, 7, 5, 2): number analyzed (Participants) | 13 | 8 | 7 | 5 | 2
  C1: AUCinf (n = 13, 8, 7, 5, 2) | 1090 (29.6) | 1080 (45.4) | 1240 (25.2) | 491 (22.7) | 1160 (7.1)
  C1: AUClast | 980 (42.5) | 1020 (109.9) | 923 (76.1) | 602 (62.2) | 865 (69.8)
  C1: AUCtau (n= 54, 55, 32, 48, 36): number analyzed (Participants) | 54 | 55 | 32 | 48 | 36
  C1: AUCtau (n= 54, 55, 32, 48, 36) | 1010 (39.8) | 1190 (35.0) | 1130 (34.9) | 689 (40.4) | 1070 (31.3)
  C3: AUC0-336h (n = 36, 49, 12, 40, 16): number analyzed (Participants) | 36 | 49 | 12 | 40 | 16
  C3: AUC0-336h (n = 36, 49, 12, 40, 16) | 1210 (36.3) | 1140 (43.8) | 1360 (45.7) | 850 (50.6) | 1290 (30.0)
  C3: AUCinf (n = 1, 1, 1, 1, 0): number analyzed (Participants) | 1 | 1 | 1 | 1 | 0
  C3: AUCinf (n = 1, 1, 1, 1, 0) | 1050 (NA) — N/A = Geometric coefficient of variation could not be calculated as there was only 1 patient | 1070 (NA) — N/A = Geometric coefficient of variation could not be calculated as there was only 1 patient | 2340 (NA) — N/A = Geometric coefficient of variation could not be calculated as there was only 1 patient | 135 (NA) — N/A = Geometric coefficient of variation could not be calculated as there was only 1 patient |
  C3: AUClast (n = 37, 51, 16, 44, 19): number analyzed (Participants) | 37 | 51 | 16 | 44 | 19
  C3: AUClast (n = 37, 51, 16, 44, 19) | 1860 (39.9) | 1650 (59.7) | 1630 (73.4) | 984 (78.0) | 1600 (88.0)
  C3: AUCtau (n= 31, 44, 7, 38, 14): number analyzed (Participants) | 31 | 44 | 7 | 38 | 14
  C3: AUCtau (n= 31, 44, 7, 38, 14) | 1940 (35.5) | 1790 (53.4) | 1920 (44.4) | 1100 (54.5) | 2120 (32.7)

8. Secondary Outcome: Phase ll: Serum Pharmacokinetic (PK) Parameter Cmax
Description: as for outcome 5
Time Frame: Predose, 1hour (h), 24h, 48h, 72h, 168h, 240h, 336h post dose (Cycle 1 & 3)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42
ug/mL
  C1 (n = 52, 58, 32, 55, 35): number analyzed (Participants) | 52 | 58 | 32 | 55 | 35
  C1 (n = 52, 58, 32, 55, 35) | 103 (37.0) | 111 (26.6) | 114 (23.6) | 79.9 (31.8) | 100 (27.3)
  C3 (n = 33, 45, 11, 39, 18): number analyzed (Participants) | 33 | 45 | 11 | 39 | 18
  C3 (n = 33, 45, 11, 39, 18) | 151 (32.0) | 141 (33.4) | 163 (34.7) | 103 (36.6) | 146 (22.6)

9. Secondary Outcome: Phase ll: Serum Pharmacokinetic (PK) Parameter Tmax
Description: as for outcome 6
Time Frame: Predose, 1hour (h), 24h, 48h, 72h, 168h, 240h, 336h post dose (Cycle 1 & 3)
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42
hour
  C1 (n= 52, 58, 32, 55, 35): number analyzed (Participants) | 52 | 58 | 32 | 55 | 35
  C1 (n= 52, 58, 32, 55, 35) | 1.58 [0.55 to 2.52] | 1.58 [1.07 to 2.9] | 1.58 [1.18 to 2.15] | 1.65 [1.00 to 3.08] | 1.55 [0.5 to 2.75]
  C3 (n = 33, 45, 11, 39, 18): number analyzed (Participants) | 33 | 45 | 11 | 39 | 18
  C3 (n = 33, 45, 11, 39, 18) | 1.6 [0.983 to 2.08] | 1.55 [1.07 to 2.22] | 1.53 [1.42 to 1.62] | 1.58 [1.33 to 2.92] | 1.57 [0 to 4.63]

10. Secondary Outcome: Phase I: Presence and/or Concentration of Anti-PDR001
Description: Assessed PDR001 anti-drug anti-body (ADA) incidence in Phase I patients - the emergence of anti-PDR001 antibodies following one or more intravenous (i.v.) infusions of PDR001. Each cycle = 28 days; End of treatment was expected to be on average 1 year after the start of study treatment.
Time Frame: 42 months
Population: Immunogenicity incidence Set: The Immunogenicity incidence set includes all subjects in FAS with a determinant baseline immunoglobulin (IG) sample and at least one determinant post-baseline IG sample.
  Treatment-induced ADA-positive was performed on ADA-positive patients only. Treatment-boosted ADA-positive was performed on ADA-positive patients only.
Measure: Number; unit: Participants
Groups:
- All Phase I q2w: Phase I dose Cohorts - All patients in Phase I who took PDR001 q2w
- All Phase I q4w: Phase I dose Cohorts - All patients in Phase I who took PDR001 q4w
- All Phase I Patients: All patients in Phase I regardless of how they took PDR001
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | All Phase I q2w | 3mg/kg q4w | 5mg/kg q4w | All Phase I q4w | All Phase I Patients
Number analyzed (Participants) | 16 | 11 | 3 | 30 | 6 | 10 | 16 | 46
Participants
  Patients with ADA-negative sample at baseline | 11 | 9 | 1 | 21 | 5 | 9 | 14 | 35
  Patients with ADA-positive sample at baseline | 5 | 2 | 2 | 9 | 1 | 1 | 2 | 11
  ADA-negative | 10 | 8 | 1 | 19 | 4 | 8 | 12 | 31
  ADA-positive (i.e., ADA incidence) | 4 | 2 | 2 | 8 | 1 | 1 | 2 | 10
  Treatment-induced ADA-positive | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 4
  Treatment-boosted ADA-positive | 3 | 1 | 2 | 6 | 0 | 0 | 0 | 6

11. Secondary Outcome: Phase II: Presence and/or Concentration of Anti-PDR001
Description: Assessed PDR001 anti-drug anti-body (ADA) incidence in Phase I patients - the emergence of anti-PDR001 antibodies following one or more intravenous (i.v.) infusions of PDR001. Each cycle = 28 days; End of treatment was expected to be on average 1 year after the start of study treatment.
  For Treatment -induced ADA-positive, Percentage was based on subjects ADA-negative at baseline.
  For Treatment-boosted ADA-positive, Percentage was based on subjects ADA-positive at baseline.
Time Frame: 42 months
Population: Immunogenicity incidence Set: The Immunogenicity incidence set includes all subjects in FAS with a determinant baseline immunoglobulin (IG) sample and at least one determinant post-baseline IG sample.
Measure: Number; unit: Participants
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w | All Phase II Patients
Number analyzed (Participants) | 52 | 54 | 33 | 46 | 31 | 216
Participants
  Patients with ADA-negative sample at baseline | 43 | 48 | 29 | 41 | 29 | 190
  Patients with ADA-positive sample at baseline | 9 | 6 | 4 | 5 | 2 | 26
  ADA-negative | 34 | 46 | 23 | 31 | 24 | 158
  ADA-positive (i.e., ADA incidence) | 11 | 4 | 7 | 12 | 6 | 40
  Treatment-induced ADA-positive | 9 | 2 | 6 | 10 | 5 | 32
  Treatment-boosted ADA-positive | 2 | 2 | 1 | 2 | 1 | 8

12. Secondary Outcome: Phase l: Overall Response Rate (ORR) as Per Investigator Based on RECIST v1.1
Description: ORR is the percentage of participants with a best overall response of complete response CR or partial response PR as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 CR = at least two determinations of CR at least 4 weeks apart before progression where confirmation required or one determination of CR prior to progression where confirmation not required.
  PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) where confirmation required or one determination of PR prior to progression where confirmation not required.
  RECIST criteria is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
Time Frame: 27 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | All Phase I q2w | 3mg/kg q4w | 5mg/kg q4w | All Phase I q4w | All Phase I Patients
Number analyzed (Participants) | 16 | 15 | 11 | 42 | 6 | 10 | 16 | 58
Percentage of participants | 0.00 [0.0 to 17.1] | 6.7 [0.3 to 27.9] | 9.1 [0.5 to 36.4] | 4.8 [0.9 to 14.2] | 0.0 [0.0 to 39.3] | 0.0 [0.0 to 25.9] | 0.0 [0.0 to 17.1] | 3.4 [0.6 to 10.5]

13. Secondary Outcome: Phase l: Disease Control Rate (DCR) as Per Investigator Based on RECIST v1.1
Description: DCR is the percentage of patients with a best overall response of CR or PR or stable disease (SD).
  CR = at least two determinations of CR at least 4 weeks apart before progression where confirmation required or one determination of CR prior to progression where confirmation not required PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) where confirmation required or one determination of PR prior to progression where confirmation not required.
  SD = at least one SD assessment (or better) > 6 weeks after randomization/start of treatment (and not qualifying for CR or PR).
  RECIST criteria is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
Time Frame: 27 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | All Phase I q2w | 3mg/kg q4w | 5mg/kg q4w | All Phase I q4w | All Phase I Patients
Number analyzed (Participants) | 16 | 15 | 11 | 42 | 6 | 10 | 16 | 58
Percentage of participants | 56.3 [33.3 to 77.3] | 46.7 [24.4 to 70.0] | 27.3 [7.9 to 56.4] | 45.2 [32.0 to 59.0] | 50.0 [15.3 to 84.7] | 20.0 [3.7 to 50.7] | 31.3 [13.2 to 54.8] | 41.4 [30.4 to 53.0]

14. Secondary Outcome: Phase l: Progression Free Survival (PFS) as Per RECIST v1.1
Description: PFS is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is per Kaplan-Meier estimates.
  RECIST criteria, published in February 2000 by an international collaboration including the European Organization for Research and Treatment of Cancer (EORTC), National Cancer Institute of the United States, and the National Cancer Institute of Canada Clinical Trials Group, is a Response evaluation criteria in solid tumors is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
  RECIST criteria is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
Time Frame: 27 months
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: Percentage of participants
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w
Number analyzed (Participants) | 16 | 15 | 6 | 11 | 10
Percentage of participants | 3.5 [1.8 to 6.5] | 1.9 [1.5 to 8.1] | 2.2 [1.7 to 5.8] | 2.7 [1.1 to 3.5] | 1.8 [1.1 to 1.8]

15. Secondary Outcome: Phase I: Duration of Response (DOR) as Per RECIST v1.1
Description: DOR is measured from the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or PD is objectively documented. CR = at least 2 determinations of CR at least 4 weeks apart before progression where confirmation required or 1 determination of CR prior to progression where confirmation not required; PR = at least 2 determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) where confirmation required or 1 determination of PR prior to progression where confirmation not required; PD =progression <= 12 weeks after randomization/start of treatment (and not qualifying for CR, PR or SD). SD = at least 1 SD assessment (or better) > 6 weeks after randomization/start of treatment (and not qualifying for CR or PR). RECIST criteria is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment
Time Frame: 27 months
Population: Full analysis set - Dose escalation
Measure: Mean (Full Range); unit: days
Arm/Group | 3mg/kg q2w | 10mg/kg q2w | All Phase I q2w | All Phase I Patients
Number analyzed (Participants) | 1 | 1 | 2 | 2
days | 261.00 [261.0 to 261.0] | 55.00 [55.0 to 55.0] | 158.00 [55.0 to 261.0] | 158.00 [55.0 to 261.0]

16. Secondary Outcome: Phase l Only: Overall Response Rate (ORR) as Per Investigator Based on Immune Related Response Criteria (irRC)
Description: ORR is the percentage of participants with a best overall response of complete response (CR) or partial response (PR) as per irRC.
  CR = at least two determinations of CR at least 4 weeks apart before progression where confirmation required or one determination of CR prior to progression where confirmation not required.
  PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) where confirmation required or one determination of PR prior to progression where confirmation not required.
  The immune-related response criteria (irRC) is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment, where the compound being evaluated is an immuno-oncology drug.
Time Frame: 27 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | All Phase I q2w | 3mg/kg q4w | 5mg/kg q4w | All Phase I q4w | All Phase I Patients
Number analyzed (Participants) | 16 | 15 | 11 | 42 | 6 | 10 | 16 | 58
Percentage of participants | 0.00 [0.0 to 17.1] | 6.7 [0.3 to 27.9] | 9.1 [0.5 to 36.4] | 4.8 [0.9 to 14.2] | 0.0 [0.0 to 39.3] | 0.0 [0.0 to 25.9] | 0.0 [0.0 to 17.1] | 3.4 [0.6 to 10.5]

17. Secondary Outcome: Phase l Only: Disease Control Rate (DCR) as Per Investigator Based on irRC
Description: DCR is the percentage of patients with a best overall response of CR or PR or stable disease (SD).
  CR = at least two determinations of CR at least 4 weeks apart before progression where confirmation required or one determination of CR prior to progression where confirmation not required PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) where confirmation required or one determination of PR prior to progression where confirmation not required.
  SD = at least one SD assessment (or better) > 6 weeks after randomization/start of treatment (and not qualifying for CR or PR).
  The immune-related response criteria (irRC) is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment, where the compound being evaluated is an immuno-oncology drug.
Time Frame: 27 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | All Phase I q2w | 3mg/kg q4w | 5mg/kg q4w | All Phase I q4w | All Phase I Patients
Number analyzed (Participants) | 16 | 15 | 11 | 42 | 6 | 10 | 16 | 58
Percentage of participants | 62.5 [39.1 to 82.2] | 53.3 [30.0 to 75.6] | 27.3 [7.9 to 56.4] | 50.0 [36.5 to 63.5] | 50.0 [15.3 to 84.7] | 30.0 [8.7 to 60.7] | 37.5 [17.8 to 60.9] | 46.6 [35.3 to 58.1]

18. Secondary Outcome: Phase l Only: Progression Free Survival (PFS) as Per irRC
Description: PFS is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is per Kaplan-Meier estimates.
  The immune-related response criteria (irRC) is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment, where the compound being evaluated is an immuno-oncology drug.
Time Frame: 27 months
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: Percentage of participants
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w
Number analyzed (Participants) | 16 | 15 | 11 | 11 | 10
Percentage of participants | 3.6 [1.8 to NA] — N/A: Model could not compute the upper limit of CI due to small sample size | 2.7 [1.5 to 8.1] | 2.2 [1.7 to 5.8] | 2.7 [1.1 to 5.2] | 1.8 [1.1 to 2.8]

19. Secondary Outcome: Phase I: Duration of Response (DOR) as Per irRC
Description: DOR: measured from time measurement criteria are met for CR or PR (whichever status is recorded first) until first date that recurrence or PD is objectively documented CR: at least 2 determinations of CR at least 4 weeks apart before progression where confirmation required or 1 determination of CR prior to progression where confirmation not required PR: at least 1 determination of PR or better at least 4 weeks apart before progression (& not qualifying for a CR) where confirmation required or 1 determination of PR prior to progression where confirmation not required PD: progression <= start of treatment (& not qualifying for CR, PR or SD) SD: at least 1 SD assessment (or better) > 6 weeks after randomization/start of treatment (& not qualifying for CR or PR) irRC is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment, where the compound being evaluated is an immuno-oncology drug
Time Frame: 61 Days
Population: Full analysis set - Dose escalation
Measure: Mean (Full Range); unit: days
Arm/Group | 3mg/kg q2w | 10mg/kg q2w | All Phase I q2w | All Phase I Patients
Number analyzed (Participants) | 1 | 1 | 2 | 2
days | 261.00 [261.0 to 261.0] | 55.00 [55.0 to 55.0] | 158.00 [55.0 to 261.0] | 158.00 [55.0 to 261.0]

20. Secondary Outcome: Phase II: Disease Control Rate (DCR) as Per Investigator Based on RECIST v1.1
Description: as for outcome 13
Time Frame: 61 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w | All Phase II Patients
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42 | 261
Percentage of participants | 49.2 [37.8 to 60.5] | 62.3 [51.0 to 72.7] | 20.0 [10.4 to 33.2] | 35.6 [25.2 to 47.1] | 31.0 [19.4 to 44.6] | 41.8 [36.6 to 47.0]

21. Secondary Outcome: Phase II: Progression Free Survival as Per Investigator Based on RECIST v1.1
Description: PFS is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is per Kaplan-Meier estimates.
  RECIST criteria, published in February 2000 by an international collaboration including the European Organization for Research and Treatment of Cancer (EORTC), National Cancer Institute of the United States, and the National Cancer Institute of Canada Clinical Trials Group, is a Response evaluation criteria in solid tumors is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
Time Frame: 61 months
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42
Percentage of participants | 2.7 [1.9 to 5.4] | 4.7 [3.5 to 5.6] | 1.7 [1.7 to 1.8] | 1.9 [1.8 to 2.1] | 1.7 [1.4 to 1.9]

22. Secondary Outcome: Phase II: Duration of Response (DOR) as Per Investigator Based on RECIST v1.1
Description: DOR is measured from the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or PD is objectively documented.
  CR = at least two determinations of CR at least 4 weeks apart before progression where confirmation required or one determination of CR prior to progression where confirmation not required PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) where confirmation required or one determination of PR prior to progression where confirmation not required.
  PD = progression <= start of treatment (and not qualifying for CR, PR or SD). SD = at least one SD assessment (or better) > 6 weeks after randomization/start of treatment (and not qualifying for CR or PR).
  RECIST criteria is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
Time Frame: 61 months
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: months
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w
Number analyzed (Participants) | 9 | 17 | 4 | 8
months | 5.6 [3.9 to 16.6] | 32.0 [11.1 to NA] — N/A = Model could not compute the upper limit of CI due to small sample size' | 10.9 [3.7 to NA] — N/A = Model could not compute the upper limit of CI due to small sample size | 22.8 [5.7 to NA] — N/A = Model could not compute the upper limit of CI due to small sample size

23. Secondary Outcome: Phase II: Overall Response Rate (ORR) as Per Investigator Based on irRC
Description: ORR is the percentage of participants with a best overall response CR or PR as per irRC.
  CR = at least two determinations of CR at least 4 weeks apart before progression where confirmation required or one determination of CR prior to progression where confirmation not required.
  PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) where confirmation required or one determination of PR prior to progression where confirmation not required.
  The immune-related response criteria (irRC) is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment, where the compound being evaluated is an immuno-oncology drug.
Time Frame: 61 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w | All Phase II Patients
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42 | 261
Percentage of participants | 18.6 [10.8 to 29.0] | 31.1 [21.5 to 42.3] | 0.0 [0.0 to 7.2] | 8.5 [3.4 to 17.0] | 23.8 [13.5 to 37.0] | 17.2 [13.5 to 21.6]

24. Secondary Outcome: Phase II: Disease Control Rate (DCR) as Per Investigator Based on irRC
Description: as for outcome 17
Time Frame: 61 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w | All Phase II Patients
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42 | 261
Percentage of participants | 55.9 [44.4 to 67.0] | 67.2 [56.0 to 77.1] | 22.5 [12.3 to 36.0] | 39.0 [28.3 to 50.5] | 35.7 [23.5 to 49.5] | 46.4 [41.1 to 51.6]

25. Secondary Outcome: Phase II: Progression Free Survival (PFS) Per irRC
Description: as for outcome 18
Time Frame: 61 months
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w
Number analyzed (Participants) | 59 | 61 | 40 | 59 | 42
Percentage of participants | 3.7 [2.6 to 7.1] | 5.4 [3.7 to 6.5] | 1.8 [1.7 to 1.8] | 2.0 [1.8 to 2.2] | 1.7 [1.4 to 1.9]

26. Secondary Outcome: Phase II: Duration of Response (DOR) Per irRC
Description: as for outcome 19
Time Frame: 61 months
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: months
Arm/Group | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w
Number analyzed (Participants) | 11 | 19 | 5 | 10
months | 5.6 [5.3 to 16.6] | 32.0 [15.6 to NA] — N/A = Model could not compute the upper limit of CI due to small sample size | 10.9 [3.7 to NA] — N/A = Model could not compute the upper limit of CI due to small sample size | 22.1 [3.8 to NA] — N/A = Model could not compute the upper limit of CI due to sparse data

27. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from the start of study treatment up to 30 days after last study treatment exposure, for a maximum duration of 114.3 weeks for Phase I part (treatment duration ranged from 2 to 110.3 weeks) and a maximum duration of 194.9 weeks for Phase II part (treatment duration ranged from 0.6 tp 190.9 weeks).
  Total deaths were collected from the start of treatment up to end of follow-up phase (approx. 70 months).
Time Frame: On treatment deaths: approx. 114.3 weeks (Phase I) & 194.9 weeks (phase II), all deaths: approx. 70 months
Population: Clinical database population: All treated patients
Measure: Number; unit: Participants
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | 3mg/kg q4w | 5mg/kg q4w | NSCLC 400 mg/q4w | Melanoma 400 mg/q4w | TNBC 400 mg/q4w | NSCLC 300 mg/q3w | ATC 400 mg/q4w
Number analyzed (Participants) | 16 | 15 | 11 | 6 | 10 | 59 | 61 | 40 | 59 | 42
Participants
  On-treatment deaths | 2 | 2 | 1 | 1 | 2 | 4 | 4 | 4 | 12 | 11
  Total deaths | 10 | 10 | 6 | 4 | 7 | 39 | 32 | 28 | 47 | 31

ADVERSE EVENTS:
Time Frame: On treatment deaths were collected from the start of study treatment up to 30 days after last study treatment exposure, for a maximum duration of 114.3 weeks for the Part I phase (treatment duration ranged from 2 to 110.3 weeks) and for a maximum duration of 194.9 weeks for the Phase II part (treatment duration ranged from 0.6 to 190.9 weeks).
Description: AE: Any sign or symptom that occurs during treatment plus 30 days post treatment.
Arm/Group | 1mg/kg q2w | 3mg/kg q2w | 10mg/kg q2w | All Phase I q2w | 3mg/kg q4w | 5mg/kg q4w | All Phase I q4w | All Phase I Patients | NSCLC 400mg/q4w | Melanoma 400mg/q4w | TNBC 400mg/q4w | NSCLC 300mg/q3w | ATC 400 mg/q4w | All Phase II Patients
All-Cause Mortality (participants affected / at risk) | 2/16 | 2/15 | 1/11 | 5/42 | 1/6 | 2/10 | 3/16 | 8/58 | 4/59 | 4/61 | 4/40 | 12/59 | 11/42 | 35/261
Serious Adverse Events (participants affected / at risk) | 9/16 | 7/15 | 4/11 | 20/42 | 2/6 | 2/10 | 4/16 | 24/58 | 27/59 | 22/61 | 18/40 | 37/59 | 22/42 | 126/261
Other Adverse Events (participants affected / at risk) | 16/16 | 15/15 | 11/11 | 42/42 | 6/6 | 10/10 | 16/16 | 58/58 | 54/59 | 55/61 | 37/40 | 56/59 | 39/42 | 241/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1mg/kg q2w (N=16) | 3mg/kg q2w (N=15) | 10mg/kg q2w (N=11) | All Phase I q2w (N=42) | 3mg/kg q4w (N=6) | 5mg/kg q4w (N=10) | All Phase I q4w (N=16) | All Phase I Patients (N=58) | NSCLC 400mg/q4w (N=59) | Melanoma 400mg/q4w (N=61) | TNBC 400mg/q4w (N=40) | NSCLC 300mg/q3w (N=59) | ATC 400 mg/q4w (N=42) | All Phase II Patients (N=261)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 4
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 3
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Complication of device insertion (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 4
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 4
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 5 | 3 | 11
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Sepsis (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 3
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 1 | 3 | 7 | 2 | 16
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 5 | 2 | 2 | 11
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 3
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lymphorrhoea (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1mg/kg q2w (N=16) | 3mg/kg q2w (N=15) | 10mg/kg q2w (N=11) | All Phase I q2w (N=42) | 3mg/kg q4w (N=6) | 5mg/kg q4w (N=10) | All Phase I q4w (N=16) | All Phase I Patients (N=58) | NSCLC 400mg/q4w (N=59) | Melanoma 400mg/q4w (N=61) | TNBC 400mg/q4w (N=40) | NSCLC 300mg/q3w (N=59) | ATC 400 mg/q4w (N=42) | All Phase II Patients (N=261)
Anaemia (Blood and lymphatic system disorders) | 5 | 7 | 2 | 14 | 1 | 3 | 4 | 18 | 16 | 13 | 6 | 8 | 11 | 54
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 1 | 6
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 6
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 1 | 5
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 1 | 2 | 1 | 13
Hypothyroidism (Endocrine disorders) | 3 | 3 | 1 | 7 | 0 | 2 | 2 | 9 | 4 | 5 | 3 | 3 | 2 | 17
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 0 | 1 | 1 | 4 | 1 | 1 | 1 | 0 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 2 | 7 | 2 | 3 | 5 | 12 | 3 | 2 | 5 | 5 | 3 | 18
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 2 | 0 | 4
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 4 | 5 | 0 | 0 | 2 | 0 | 0 | 2
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 0 | 10 | 2 | 0 | 2 | 12 | 8 | 7 | 9 | 9 | 5 | 38
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 1 | 14 | 0 | 3 | 3 | 17 | 8 | 8 | 1 | 12 | 8 | 37
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 1 | 5 | 0 | 1 | 1 | 6 | 3 | 3 | 1 | 0 | 3 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 3 | 0 | 1 | 1 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 5 | 8
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 4 | 3 | 14 | 3 | 4 | 7 | 21 | 9 | 6 | 13 | 15 | 2 | 45
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 6
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1 | 3 | 10 | 2 | 2 | 4 | 14 | 8 | 8 | 5 | 8 | 3 | 32
Asthenia (General disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 12 | 8 | 4 | 12 | 8 | 44
Chills (General disorders) | 2 | 1 | 1 | 4 | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 2 | 1 | 6
Face oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 10 | 3 | 2 | 15 | 2 | 5 | 7 | 22 | 11 | 12 | 13 | 12 | 6 | 54
Inflammation (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2
Malaise (General disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 4
Non-cardiac chest pain (General disorders) | 1 | 2 | 1 | 4 | 0 | 1 | 1 | 5 | 2 | 3 | 2 | 8 | 0 | 15
Oedema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 2 | 5 | 0 | 1 | 1 | 6 | 5 | 3 | 5 | 4 | 7 | 24
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 5
Peripheral swelling (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 2 | 2 | 1 | 5 | 0 | 1 | 1 | 6 | 9 | 9 | 3 | 11 | 9 | 41
Swelling face (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 6
Laryngitis bacterial (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 2 | 6
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 3
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 3 | 3 | 10
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 8 | 0 | 2 | 0 | 13
Urinary tract infection (Infections and infestations) | 1 | 3 | 0 | 4 | 0 | 0 | 0 | 4 | 2 | 2 | 1 | 2 | 0 | 7
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3 | 1 | 0 | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 3 | 2 | 7 | 5 | 5 | 3 | 22
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2 | 5 | 0 | 1 | 1 | 6 | 3 | 7 | 8 | 5 | 2 | 25
Bacterial test positive (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 0 | 5 | 0 | 0 | 0 | 5 | 2 | 2 | 6 | 3 | 1 | 14
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 1 | 5
Blood creatinine decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 3 | 1 | 4 | 1 | 4 | 0 | 10
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 1 | 8
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 5
Transaminases increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 4 | 2 | 1 | 7 | 1 | 3 | 4 | 11 | 6 | 5 | 2 | 9 | 2 | 24
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 4
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 3 | 9 | 2 | 2 | 4 | 13 | 18 | 13 | 7 | 17 | 5 | 60
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3 | 2 | 0 | 2 | 5 | 0 | 0 | 0 | 1 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3 | 1 | 0 | 1 | 4 | 4 | 0 | 0 | 2 | 3 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 4 | 0 | 0 | 0 | 4 | 1 | 4 | 1 | 3 | 2 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 2 | 3 | 4 | 2 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 5 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4 | 1 | 0 | 1 | 5 | 2 | 3 | 2 | 6 | 4 | 17
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 3 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 6 | 0 | 1 | 1 | 7 | 2 | 3 | 4 | 2 | 3 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3 | 0 | 1 | 1 | 4 | 3 | 4 | 1 | 1 | 2 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 4 | 1 | 2 | 3 | 7 | 8 | 7 | 0 | 6 | 6 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4 | 1 | 0 | 1 | 5 | 8 | 1 | 3 | 10 | 5 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 0 | 8
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 3 | 1 | 2 | 1 | 0 | 0 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 1 | 0 | 1 | 4 | 1 | 4 | 3 | 1 | 1 | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 2 | 2 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3 | 0 | 1 | 1 | 4 | 5 | 1 | 1 | 9 | 3 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3 | 2 | 0 | 2 | 5 | 4 | 4 | 1 | 1 | 3 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 3 | 4 | 10
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 4 | 1 | 1 | 2 | 6 | 1 | 4 | 3 | 4 | 0 | 12
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 5 | 0 | 8
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 3 | 10
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 6 | 0 | 10 | 0 | 0 | 0 | 10 | 1 | 5 | 4 | 10 | 3 | 23
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 4 | 1 | 6 | 1 | 3 | 4 | 10 | 4 | 4 | 2 | 7 | 5 | 22
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 6
Paralysis (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 3
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 2 | 8
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 1 | 2 | 2 | 7
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 4 | 5 | 2 | 6 | 4 | 5 | 2 | 19
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 5
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 7 | 0 | 3 | 3 | 10 | 13 | 8 | 10 | 20 | 6 | 57
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 2 | 14 | 0 | 4 | 4 | 18 | 17 | 1 | 10 | 18 | 9 | 55
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 4 | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 4 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 5 | 0 | 2 | 2 | 7 | 3 | 1 | 4 | 3 | 1 | 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 6 | 1 | 3 | 2 | 3 | 15
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 4
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 9 | 0 | 0 | 0 | 9 | 7 | 8 | 4 | 3 | 5 | 27
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 5 | 6 | 3 | 3 | 3 | 20
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 3 | 2 | 3 | 0 | 1 | 1 | 7
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 1 | 11
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 3
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 3
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 3

LIMITATIONS AND CAVEATS:
Although the study had 2 'arms', the phase I part of the study had 5 dosing cohorts and the phase ll part had 5 treatment groups for a total of 10 reporting groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT02404441/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT02404441/SAP_001.pdf